CLINICAL TRIAL: NCT04823676
Title: Efficacy and Safety of a Probiotic Composition as Adjunct Treatment in the Comprehensive Management of Metabolism-Associated Hepatic Steatosis in Adults
Brief Title: Efficacy and Safety of a Probiotic Composition as Adjunct in MAFL Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABB-MAFL21A
Record Dates: First submitted 2021-03-15; First posted 2021-04-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Non Alcoholic Fatty Liver
Keywords: NAFL; MAFL
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active and placebo capsules are indistinguishable in form, color and taste, and provided in coded boxes. List containing the correspondence between codes and treatment group assignment is prepared by a pharmacist not participating in the study and kept in a sealed envelope until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic composition (Active Comparator): A capsule containing a mix of probiotic strains (1.5 x 10^9 CFU/capsule ) administered once daily for 4 months
  Interventions: Dietary Supplement: Probiotic composition
- Placebo (Placebo Comparator): A capsule containing placebo administered once daily for 4 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic composition — Mixture of two Lactoplantibacillus plantarum strains (formerly Lactobacillus plantarum) and one Levilactobacillus brevis strain (formerly Lactobacillus brevis), in a maltodextrin carrier (E1400)
  Arms: Probiotic composition
Other: Placebo — Maltodextrin (E1400, qs)
  Arms: Placebo

SUMMARY:
Some studies have shown beneficial results with probiotics on hepatic function of subjects with fatty liver, but significant variability has been noted among probiotic formulations. This study aims at providing a comprehensive characterization of the effect of a particular probiotic formula in hepatic function of said subjects.

DETAILED DESCRIPTION:
Some studies have shown beneficial results with probiotics on hepatic function of subjects with Non-Alcoholic Fatty Liver (NAFL) also known as Metabolism-Associated Fatty Liver (MAFL). However, meta-analyses have found significant variability among probiotic formulations. In fact, many probiotic properties are thought to be strain-specific.

This study aims at providing a comprehensive characterization of a particular probiotic formula containing Lactoplantibacillus plantarum (formerly Lactobacillus plantarum) and Levilactobacillus brevis (formerly Lactobacillus brevis) in hepatic function of individuals with NAFL. The study will assess hepatic stiffness via transient elastography (Fibroscan), hepatic function via liver enzymes in serum (ALT, AST, GGT) and liver-specific inflammation via cytokeratin18 in serum, as well as some general metabolic and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hepatic Steatosis associated with Metabolism (MAFL, also known as Non-Alcoholic Fatty Liver or NAFL) with Controlled Attenuation Parameter (CAP) value of > 269 dB / m when evaluated by Fibroscan transient elastography
* Alanine aminotransferase (ALT) levels at least 35% above the upper limit of reference values
* BMI between 25 and 40 kg / m2
* Signing of the informed consent and understanding of the procedures to be carried out
* Not willing to change their current dietary habits (hypercaloric and hyperlipemic)

Exclusion Criteria:

* Treatment of NAFL or NASH (Non-Alcoholic Steato-Hepatitis) for at least 3 months prior to the study, with high dose vitamin E (≥200 mg / day), high dose omega-3 (≥500 mg / day), pioglitazone, bile acid sequestrants, statins, GLP-1 agonists, and / or DPP4 inhibitors ("gliptins"), and not having shown a significant biochemical and ultrasonographic improvement
* History of chronic alcohol or drug abuse
* Diagnosis of infectious hepatitis or HIV infection
* Diagnosis of hemochromatosis
* Celiac disease, inflammatory bowel disease, chronic or recurrent diarrhea
* Chronic use of laxatives.
* Pancreatic failure, thyroid dysfunction, severe liver disease, biliary dysfunction (including cholecystectomy and blood bilirubin abnormalities)
* Uncontrolled diabetes or hypertriglyceridemia greater than 500mg / dL
* History of regular use (> 3 days) of oral or parenteral antibiotics one month prior to the study
* Current use of systemic corticosteroids, androgens, clopidogrel, digoxin, acenocoumarol, warfarin, phenytoin, topiramate, lithium, tricyclic antidepressants, monoamine oxidase inhibitors, second generation antipsychotics, amiodarone, tamoxifen, and/or diltiazem.
* Intake of other probiotics, plant-derived sterols, beta-glucans, red rice yeast (Monascus purpureus), or milk thistle extract (Silybum marianum) or its active ingredients (silymarin, silybin) on a regular basis (> 7 days) in the 15 days prior to entering the study.
* History of angina or cardiovascular events, cancer, or immunosuppression
* Chronic, moderate-to-heavy smoking (> 5 cigarettes a day)
* History of gastro-intestinal surgery in the previous year.
* Debilitating diseases (advanced liver or kidney disease, severe depression, psychotic symptoms, neurological diseases).
* Current pregnancy (positive urine test), or planning to become pregnant during the course of the study.
* Breastfeeding at the time of eligibility assessment
* Subjects having participated in a clinical study within 1 month prior to eligibility assessment
* Current use of 4 or more concomitant medications of any type

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Change in alanine amino transferase (ALT) | change month 2 from baseline
  Change in serum levels (international units/L) of alanine amino transferase (ALT) across the study. Sample obtained through blood sampling
Change in alanine amino transferase (ALT) | change month 4 from baseline
  Change in serum levels (international units/L) of alanine amino transferase (ALT) across the study. Sample obtained through blood sampling

SECONDARY OUTCOMES:
Change in hepatic steatosis | change month 2 from baseline
  Change in the severity of the degree of hepatic steatosis measured by transient elastography with controlled attenuation parameter (Fibroscan CAP®)
Change in hepatic steatosis | change month 4 from baseline
  Change in the severity of the degree of hepatic steatosis measured by transient elastography with controlled attenuation parameter (Fibroscan CAP®)
Change in Fibroscan-AST score | change month 2 from baseline
  Change in the values of the Fibroscan-AST score (FAST, ranging 0-1), where higher values indicate a worse condition
Change in Fibroscan-AST score | change month 4 from baseline
  Change in the values of the Fibroscan-AST score (FAST, ranging 0-1), where higher values indicate a worse condition
Change in Fatty Liver Index | change month 2 from baseline
  Change in the values of the Fatty Liver Index (FLI, ranging 0-100), where higher values indicate a worse condition
Change in Fatty Liver Index | change month 4 from baseline
  Change in the values of the Fatty Liver Index (FLI, ranging 0-100), where higher values indicate a worse condition
Change in Hepatic Steatosis Index | change month 2 from baseline
  Change in the values of the Hepatic Steatosis Index (HSI, ranging 0-100), where higher values indicate a worse condition
Change in Hepatic Steatosis Index | change month 4 from baseline
  Change in the values of the Hepatic Steatosis Index (HSI, ranging 0-100), where higher values indicate a worse condition
Change in Cholesterol | change month 2 from baseline
  Change in LDL cholesterol, oxidized LDL-cholesterol, HDL-cholesterol, non-HDL cholesterol, total cholesterol. Sample obtained through blood sampling.
Change in Cholesterol | change month 4 from baseline
  Change in LDL cholesterol, oxidized LDL-cholesterol, HDL-cholesterol, non-HDL cholesterol, total cholesterol. Sample obtained through blood sampling.
Change in leptin serum parameters | change month 2 from baseline
  Change in leptin. Sample obtained through blood sampling.
Change in leptin serum parameters | change month 4 from baseline
  Change in leptin. Sample obtained through blood sampling.
Change in adiponectin serum parameters | change month 2 from baseline
  Change in adiponectin. Sample obtained through blood sampling.
Change in adiponectin serum parameters | change month 4 from baseline
  Change in adiponectin. Sample obtained through blood sampling.
Change in HOMA serum parameters | change month 2 from baseline
  Change in HOMA (Homeostatic Model Assessment). Sample obtained through blood sampling.
Change in HOMA serum parameters | change month 4 from baseline
  Change in HOMA (Homeostatic Model Assessment). Sample obtained through blood sampling.
Change in glucose serum parameters | change month 2 from baseline
  Change in glucose. Sample obtained through blood sampling.
Change in glucose serum parameters | change month 4 from baseline
  Change in glucose. Sample obtained through blood sampling.
Change in glycosylated hemoglobin serum parameters | change month 2 from baseline
  Change in glycosylated hemoglobin (Hb1Ac). Sample obtained through blood sampling.
Change in glycosylated hemoglobin serum parameters | change month 4 from baseline
  Change in glycosylated hemoglobin (Hb1Ac). Sample obtained through blood sampling.
Change in insulin serum parameters | change month 2 from baseline
  Change in insulin. Sample obtained through blood sampling.
Change in insulin serum parameters | change month 4 from baseline
  Change in insulin. Sample obtained through blood sampling.
Change in Triglycerides serum parameters | change month 2 from baseline
  Change in Triglycerides. Sample obtained through blood sampling.
Change in Triglycerides serum parameters | change month 4 from baseline
  Change in Triglycerides. Sample obtained through blood sampling.
Change in ferritin serum parameters | change month 2 from baseline
  Change in ferritin. Samples obtained through blood sampling
Change in ferritin serum parameters | change month 4 from baseline
  Change in ferritin. Samples obtained through blood sampling
Change in C-reactive protein serum parameters | change month 2 from baseline
  Change in ferritin. Samples obtained through blood sampling
Change in C-reactive protein serum parameters | change month 4 from baseline
  Change in ferritin. Samples obtained through blood sampling
Change in IL-1beta serum parameters | change month 2 from baseline
  Change in IL-1beta. Samples obtained through blood sampling
Change in IL-1beta serum parameters | change month 4 from baseline
  Change in IL-1beta. Samples obtained through blood sampling
Change in TNF-alpha serum parameters | change month 2 from baseline
  Change in TNF-alpha. Samples obtained through blood sampling
Change in TNF-alpha serum parameters | change month 4 from baseline
  Change in TNF-alpha. Samples obtained through blood sampling
Change in Cytokeratin-18 serum parameters | change month 2 from baseline
  Change in Cytokeratin-18. Samples obtained through blood sampling
Change in Cytokeratin-18 serum parameters | change month 4 from baseline
  Change in Cytokeratin-18. Samples obtained through blood sampling
Change in IL-17 serum parameters | change month 4 from baseline
  Change in IL-17. Samples obtained through blood sampling
Change in IL-17 serum parameters | change month 2 from baseline
  Change in IL-17. Samples obtained through blood sampling
Intestinal microbiota composition | change month 4 from baseline
  Change in alpha and beta diversity of the gut microbiota as assessed by 16S bacterial gene analysis
Change in fat values | change month 2 from baseline
  Change in the values of total body fat and visceral fat evaluated by impedance measurement
Change in fat values | change month 4 from baseline
  Change in the values of total body fat and visceral fat evaluated by impedance measurement
Change in waist values | change month 2 from baseline
  Change in the values of waist circumference evaluated by impedance measurement
Change in waist values | change month 4 from baseline
  Change in the values of waist circumference evaluated by impedance measurement
Change in waist / height index | change month 2 from baseline
  Change in the values of waist / height index, evaluated by impedance measurement
Change in waist / height index | change month 4 from baseline
  Change in the values of waist / height index, evaluated by impedance measurement
Change in hip circumference values | change month 2 from baseline
  Change in the hip circumference evaluated by impedance measurement
Change in hip circumference values | change month 4 from baseline
  Change in the hip circumference evaluated by impedance measurement
Change in BMI values | change month 2 from baseline
  Change in the values of Body Mass Index (BMI) evaluated by impedance measurement
Change in BMI values | change month 4 from baseline
  Change in the values of Body Mass Index (BMI) evaluated by impedance measurement
Adverse events | Throughout study completion, an average of 4 months
  Frequency of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma YY, Li L, Yu CH, Shen Z, Chen LH, Li YM. Effects of probiotics on nonalcoholic fatty liver disease: a meta-analysis. World J Gastroenterol. 2013 Oct 28;19(40):6911-8. doi: 10.3748/wjg.v19.i40.6911. PMID 24187469
- [Result] Loman BR, Hernandez-Saavedra D, An R, Rector RS. Prebiotic and probiotic treatment of nonalcoholic fatty liver disease: a systematic review and meta-analysis. Nutr Rev. 2018 Nov 1;76(11):822-839. doi: 10.1093/nutrit/nuy031. PMID 30113661
- [Result] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Result] Bedogni G, Bellentani S, Miglioli L, Masutti F, Passalacqua M, Castiglione A, Tiribelli C. The Fatty Liver Index: a simple and accurate predictor of hepatic steatosis in the general population. BMC Gastroenterol. 2006 Nov 2;6:33. doi: 10.1186/1471-230X-6-33. PMID 17081293
- [Result] Lee JH, Kim D, Kim HJ, Lee CH, Yang JI, Kim W, Kim YJ, Yoon JH, Cho SH, Sung MW, Lee HS. Hepatic steatosis index: a simple screening tool reflecting nonalcoholic fatty liver disease. Dig Liver Dis. 2010 Jul;42(7):503-8. doi: 10.1016/j.dld.2009.08.002. Epub 2009 Sep 18. PMID 19766548
- [Result] Newsome PN, Sasso M, Deeks JJ, Paredes A, Boursier J, Chan WK, Yilmaz Y, Czernichow S, Zheng MH, Wong VW, Allison M, Tsochatzis E, Anstee QM, Sheridan DA, Eddowes PJ, Guha IN, Cobbold JF, Paradis V, Bedossa P, Miette V, Fournier-Poizat C, Sandrin L, Harrison SA. FibroScan-AST (FAST) score for the non-invasive identification of patients with non-alcoholic steatohepatitis with significant activity and fibrosis: a prospective derivation and global validation study. Lancet Gastroenterol Hepatol. 2020 Apr;5(4):362-373. doi: 10.1016/S2468-1253(19)30383-8. Epub 2020 Feb 3. PMID 32027858
- [Derived] Aghara H, Patel M, Chadha P, Parwani K, Chaturvedi R, Mandal P. Unraveling the Gut-Liver-Brain Axis: Microbiome, Inflammation, and Emerging Therapeutic Approaches. Mediators Inflamm. 2025 Jun 18;2025:6733477. doi: 10.1155/mi/6733477. eCollection 2025. PMID 40568349